CLINICAL TRIAL: NCT06333106
Title: PoCUS Diagnostic Accuracy for Fecal Impaction in the Emergency Department: A Prospective Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Grand Hôpital de Charleroi (Other); Jolimont (Unknown); University of Liege (Other); Clinique Saint Pierre Ottignies (Other); Clinique Saint-Jean, Bruxelles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FICUS - 2024/16FEV/077
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Fecal Impaction of Colon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient suspected to suffer from fecal impaction (Other): Any patients aged 75 years or older coming to the ED and for whom the emergency physician suspects fecal impaction.
  Interventions: Other: POCUS diagnostic value

INTERVENTIONS:
Other: POCUS diagnostic value — Evaluation of the diagnostic value of clinical ultrasound in the diagnosis of fecal impaction in the emergency room

SUMMARY:
Many medical and paramedical specialties regularly use point-of-care ultrasound (PoCUS) in clinical practice. The diagnosis of fecal impaction is quite common in the elderly living in nursing homes with a prevalence of 47.3%. Fecal impaction remains a major source of morbidity, while its etiology is often multifactorial and its diagnosis challenging. Current recommendations for the diagnosis of fecal impaction support the use of plain abdominal x-rays. PoCUS is a non-irradiating procedure and a clinical diagnostic tool that can be used in a variety of ways during abdominal examinations. Most scientific societies encourage the use of PoCUS to respond to a specific clinical question rather than to provide a diagnosis, which is usually confirmed by conventional ultrasound. However, the combination of physical examination and PoCUS may improve the diagnostic approach. This multicentric prospective study protocol aims to evaluate the diagnostic accuracy of PoCUS in patients aged 75 years or older with suspected fecal impaction in the emergency department compared with plain abdominal x-ray (or abdominal CT scan if required as part of the emergency department investigations).

DETAILED DESCRIPTION:
Background Many medical specialties and paramedical fields are increasingly using point-of-care ultrasound (PoCUS). PoCUS is a pillar of clinical evaluation along with inspection, palpation, percussion, and auscultation, and it has become essential in daily clinical practice, as it enhances differential diagnosis. In a position statement published in 2015, the American Academy of Emergency Medicine followed by the European Federation of Societies for Ultrasound in Medicine and Biology in 2016 recommended the inclusion of PoCUS in the curricula of medical schools to improve the learning of core concepts and enhance students' understanding of physical examinations. The integration of PoCUS into clinical examination raises the issue of PoCUS diagnostic accuracy.

In everyday practice, fecal impaction is defined as the accumulation of hard fecal matter in the rectum and colon, with the absence of spontaneous evacuation. Its annual prevalence is estimated at 47.3% in nursing homes, affecting approximately 70% of nursing home patients. Furthermore, 42% of patients admitted to geriatric services suffer from fecal impaction.

In the United States, 21.9% of patients admitted to the emergency department (ED) with fecal impaction died in hospital, and severe morbidity was identified in 40.6% of patients. Over 90% of the patients with fecal impaction who visited the ED subsequently required hospitalization. In 2011, there were 42,000 ED visits in the US for fecal impaction, with patients aged over 65 being the most affected.

It is widely known that the incidence of fecal impaction increases with age and impairs quality of life in patients over 65 years of age. This common problem is often undiagnosed and thus frequently left untreated, whereas its prompt identification and treatment minimize the risk of complications. The most frequent symptoms are false diarrhea, fecal incontinence, behavioral disorders (agitation, delirium), loss of appetite, nausea, vomiting, abdominal pain, and electrolyte disorders. The site of impaction is most often rectal in 66.4% of cases. Fecal impaction is the most frequent cause of diarrhea in the elderly, with an incidence of 55%. Currently, in the ED, fecal impaction is diagnosed by plain abdominal X-rays or abdominal computed tomography (CT) scans if required as part of the ED investigations.

PoCUS is a valuable tool for investigating suspected fecal impaction, as it can guide the investigator to make a rapid diagnosis, thus leading to its rapid management. To analyze the presence of fecal impaction using PoCUS, the patient should be supine and comfortable. In the case of fecal retention in the rectal lumen, ultrasound waves are reflected from the surface of the contents at a depth deeper than the bladder (anechoic area), with a hyperechoic area with a half-moon shape being depicted in the transverse ultrasound image. In addition, with hard stool accumulation, an acoustic shadow appears in the transverse ultrasound image of the crescent-shaped hyperechoic area. By contrast, in the absence of fecal retention or gas in the rectal lumen, no obvious hyperechoic area is depicted. In the transverse ultrasound image, a circumferential hypoechoic area may be observed as an empty intestine.

The main objective of this study is to evaluate the contribution of PoCUS to the clinical examination of patients coming to the ED with clinical suspicion of fecal impaction.

Trial design This study is an interventional multicentric prospective study aiming to evaluate PoCUS diagnosis accuracy in patients aged 75 years or older presenting to the ED with suspected fecal impaction while taking a plain abdominal x-ray (or abdominal CT scan if required for the ED investigations) as the reference diagnostic investigation.

Inclusion process The emergency physician in charge of the eligible patients with suspected fecal impaction will advise the investigator before ordering a plain x-ray.

The investigator will assess the patient's eligibility, explain the study, and obtain signed informed consent. She or he will then verify the inclusion and exclusion criteria and initiate the study process.

Intervention process The investigator is independent of the patient medical management. She or he will perform an abdominal ultrasound in search of fecal impaction. PoCUS images will be recorded according to the procedures of the study centers and their capacities in terms of the ultrasound equipment.

The investigator will complete a case report form (CRF) stipulating the presence or absence of fecal impaction (Appendix 1). The diagnosis of fecal impaction will be made based on a plain abdominal x-ray (or abdominal CT scan if required as part of the ED investigations).

In the case of a positive x-ray, the emergency physician will perform a digital rectal examination to determine the consistency of the fecal impaction (hard or soft) and initiate the appropriate treatment.

Evaluation process A research associate will record the anonymous CRF data on a dedicated computerized database (REDCAP). Based on the recorded data, the diagnostic accuracy of PoCUS for fecal impaction will be determined.

Sample size The sample includes patients aged 75 years or over presenting to the ED with suspected fecal impaction. The diagnostic value of clinical or radiological ultrasound for fecal impaction is not precisely known. Based on a 42% prevalence of fecal impaction in elderly patients, a sample of 247 patients is required to obtain a 95% confidence interval for an expected sensitivity of 95%, assuming an attrition rate of 10%.

Statistical method The software IBM SPSS statistics 26.0 (SPSS Inc., Chicago, IL, USA) will be used to analyze the data. Continuous variables describing the study population will be detailed using medians, standard deviations, and minimum and maximum values. Discrete variables will be reported by category as numbers and percentages. The χ² test of independence will be used to compare discrete variables. The Wilcoxon-Mann-Whitney test will be used to compare continuous variables. The significance level corresponds to a p-value of 0.05 or less. The 95% confidence intervals will be calculated using the mid-p exact value.

Data management Data collection All the data relating to this study will be collected on paper CRF by the study investigator. Collected data will concern the clinical situation, patient characteristics, test results, and diagnostic approach associated with the coefficients of certainty of the physicians in charge as well as any questions relating to the bedside PoCUS. Any missing data will be collected from the medical file by the inclusion center's principal investigator, coordinating investigator, or research associates. Patients will initially be identified on the CRF by their last name, first name, date of birth, file number from the institution where they were included, and an identification number of the study.

This identification number will be comprised of a reference for the inclusion center and participant number. After the principal investigators or research associates complete the collection of missing data, patients will henceforth only be identified by their study identification number to anonymize the data. Data will be recorded on REDCAP.

Data access A list of correspondence between the study identification number and the other identifying data will be kept under the responsibility of the project promoter. This list is kept for the statutory period of time provided for this type of research. The protection of patients' personal data will be guaranteed by the European General Data Protection Regulation of April 27, 2016 (in application since May 25, 2018), the Belgian Law of July 30, 2018, on privacy protection with regard to the processing of personal data, and the Belgian Law of August 22, 2002, on patient rights.

Certified good clinical practice will be used with a compliant electronic data management system. The system is connected to the clinical center database management system, thus restricting access to authorized users. This distinguishes between users and guarantees data safety.

Any individual with direct access to the data will take all the necessary precautions to ensure the confidentiality of the information relating to participants included in the study, particularly regarding their identity and results. Any individual with direct access to data will be subject to professional secrecy. They will undertake to never divulge the confidential information relating to the study participants and to guarantee the anonymization of the data before transferring it to the database manager and biostatistician. Any data disclosure required by the law or applicable regulations will be done if necessary.

Data storage After completing the data collection and anonymization, the data will be added to a file (SPSS 26.0) with access restricted by a password. This document will be owned by the project promoter represented by the study coordinator. This person ensures that the documents and data relating to the research are kept for 20 years in accordance with the applicable regulations. Coordinating investigators are responsible for keeping the essential study documents at the research site. If they leave the institution, they will delegate this responsibility to the project promoter in writing.

Ethics Written documentation explaining the PoCUS procedure and the risks or benefits of undergoing PoCUS will be given to all participants. They will also receive an explanation of data protection.

Ultrasound technology does not put participants at risk during abdominal ultrasound. Indeed, physicians are required to observe the ALARA (as low as reasonably achievable) principle during clinical examinations. Signed written consent to participate in this study will be collected for each participant as recommended by the Additional Protocol to the Convention on Human Rights and Biomedicine concerning Biomedical Research as well as by the Council of Europe's Steering Committee on Bioethics.

A study file including this protocol, a research summary, and the CRF will be submitted to the ethics committees of each participating center. The research protocol will only begin if a favorable opinion is granted by the local ethics committees as well as the ethics committee of the main center. Any substantial changes made to the study file must be approved by the study promoter. Before making any changes, all the ethics committees will need to give their approval. The project promoter will communicate the study end date to the ethics committees within a delay of 90 days. This date will correspond to the date of the last inclusion or, if appropriate, to the theoretical end date of the study in this protocol. If the inclusion number is not reached within 6 months, an extension request will be added to the protocol.

Compensation No compensation is given to the participants of this study. Adverse event An adverse event is any untoward medical occurrence in a patient, including the exacerbation of an existing condition that is not necessarily related to the study itself. Any incidental findings using PoCUS will be reported, and information will be forwarded to patients under medical confidentiality. The family physician will also be notified by telephone and in a consultation letter from the ED. All the results will be recorded confidentially in the patient's medical file. The reasons for losing participants to follow-up will also be mentioned.

This is a clinical study. PoCUS is a non-invasive procedure for which no risks have been reported in the current literature. In this study, patient management will always take priority over performing PoCUS.

Insurance Regarding the Belgian law of May 7, 2004, the project promoter will take out insurance to cover any risk incurred by the study participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients 75 years or older
* Patient for whom the clinician in charge indicates that an abdominal x-ray should be performed to check for the presence of a fecal impaction
* Informed consent, read and signed by the patient or their legal representative

Exclusion Criteria:

* Patient or legal representative not understanding one of the consent languages (French, Dutch and English)
* Reasons making suprapubic ultrasound impossible

Ages: 75 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 247 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of the diagnostic value of clinical ultrasound in the diagnosis of fecal impaction in the emergency room | 2 hours
  Sensitivity and specificity of PoCUS in the diagnosis of fecal impaction compared to abdominal radiography (or abdominal CT) as a diagnostic reference tool with likelihood ratios and positive and negative predictive values.

SECONDARY OUTCOMES:
Influence of BMI on the diagnosis of fecal impaction at PoCUS | 2 hours
  Proportion test
Influence of bladder repletion on the diagnosis of fecal impaction using PoCUS | 2 hours
  Proportion test
Influence of patient echogenicity on the diagnosis of fecal impaction using PoCUS | 2 hours
  Proportion test

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Penaloza, MD, PhD, Study Director — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (6):
- Belgium (6):
  - Clinique Saint-Jean, Bruxelles, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Grand Hôpital de Charleroi, Charleroi
  - Jolimont, La Louvière
  - Université de Liège, Liège
  - Clinique Saint Pierre Ottignies, Ottignies-Louvain-la-Neuve

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meadley B, Olaussen A, Delorenzo A, Roder N, Martin C, St Clair T, Burns A, Stam E, Williams B. Educational standards for training paramedics in ultrasound: a scoping review. BMC Emerg Med. 2017 Jun 17;17(1):18. doi: 10.1186/s12873-017-0131-8. PMID 28623905
- [Background] Soucy ZP, Mills LD. American Academy of Emergency Medicine Position Statement: Ultrasound Should Be Integrated into Undergraduate Medical Education Curriculum. J Emerg Med. 2015 Jul;49(1):89-90. doi: 10.1016/j.jemermed.2014.12.092. Epub 2015 Apr 29. No abstract available. PMID 25934381
- [Background] Cantisani V, Dietrich CF, Badea R, Dudea S, Prosch H, Cerezo E, Nuernberg D, Serra AL, Sidhu PS, Radzina M, Piscaglia F, Bachmann Nielsen M, Ewertsen C, Saftoiu A, Calliada F, Gilja OH. EFSUMB Statement on Medical Student Education in Ultrasound [long version]. Ultrasound Int Open. 2016 Mar;2(1):E2-7. doi: 10.1055/s-0035-1569413. PMID 27689163
- [Background] Nicholas E, Ly AA, Prince AM, Klawitter PF, Gaskin K, Prince LA. The Current Status of Ultrasound Education in United States Medical Schools. J Ultrasound Med. 2021 Nov;40(11):2459-2465. doi: 10.1002/jum.15633. Epub 2021 Jan 15. PMID 33448471
- [Background] Prosch H, Radzina M, Dietrich CF, Nielsen MB, Baumann S, Ewertsen C, Jenssen C, Kabaalioglu A, Kosiak W, Kratzer W, Lim A, Popescu A, Mitkov V, Schiavone C, Wohlin M, Wustner M, Cantisani V. Ultrasound Curricula of Student Education in Europe: Summary of the Experience. Ultrasound Int Open. 2020 Jun;6(1):E25-E33. doi: 10.1055/a-1183-3009. Epub 2020 Aug 31. PMID 32885138
- [Background] Atkinson P, Bowra J, Lambert M, Lamprecht H, Noble V, Jarman B. International Federation for Emergency Medicine point of care ultrasound curriculum. CJEM. 2015 Mar;17(2):161-70. doi: 10.1017/cem.2015.8. PMID 26052968
- [Background] Hayward SA, Janssen J. Use of thoracic ultrasound by physiotherapists: a scoping review of the literature. Physiotherapy. 2018 Dec;104(4):367-375. doi: 10.1016/j.physio.2018.01.001. Epub 2018 Feb 2. PMID 29958691
- [Background] Rey E, Barcelo M, Jimenez Cebrian MJ, Alvarez-Sanchez A, Diaz-Rubio M, Rocha AL. A nation-wide study of prevalence and risk factors for fecal impaction in nursing homes. PLoS One. 2014 Aug 22;9(8):e105281. doi: 10.1371/journal.pone.0105281. eCollection 2014. PMID 25148393
- [Background] Barcelo M, Jimenez-Cebrian MJ, Diaz-Rubio M, Rocha AL, Rey E. Validation of a questionnaire for assessing fecal impaction in the elderly: impact of cognitive impairment, and using a proxy. BMC Geriatr. 2013 Mar 7;13:24. doi: 10.1186/1471-2318-13-24. PMID 23496919
- [Background] Sommers T, Petersen T, Singh P, Rangan V, Hirsch W, Katon J, Ballou S, Cheng V, Friedlander D, Nee J, Lembo A, Iturrino J. Significant Morbidity and Mortality Associated with Fecal Impaction in Patients Who Present to the Emergency Department. Dig Dis Sci. 2019 May;64(5):1320-1327. doi: 10.1007/s10620-018-5394-8. Epub 2018 Dec 8. PMID 30535766
- [Background] Corban C, Sommers T, Sengupta N, Jones M, Cheng V, Friedlander E, Bollom A, Lembo A. Fecal Impaction in the Emergency Department: An Analysis of Frequency and Associated Charges in 2011. J Clin Gastroenterol. 2016 Aug;50(7):572-7. doi: 10.1097/MCG.0000000000000458. PMID 26669560
- [Background] Kinnunen O, Jauhonen P, Salokannel J, Kivela SL. Diarrhea and fecal impaction in elderly long-stay patients. Z Gerontol. 1989 Nov-Dec;22(6):321-3. PMID 2623935
- [Background] Matsumoto M, Misawa N, Tsuda M, Manabe N, Kessoku T, Tamai N, Kawamoto A, Sugama J, Tanaka H, Kato M, Haruma K, Sanada H, Nakajima A. Expert Consensus Document: Diagnosis for Chronic Constipation with Faecal Retention in the Rectum Using Ultrasonography. Diagnostics (Basel). 2022 Jan 25;12(2):300. doi: 10.3390/diagnostics12020300. PMID 35204390
- [Background] Miller DL, Abo A, Abramowicz JS, Bigelow TA, Dalecki D, Dickman E, Donlon J, Harris G, Nomura J. Diagnostic Ultrasound Safety Review for Point-of-Care Ultrasound Practitioners. J Ultrasound Med. 2020 Jun;39(6):1069-1084. doi: 10.1002/jum.15202. Epub 2019 Dec 23. PMID 31868252
- [Background] Booth TC, Jackson A, Wardlaw JM, Taylor SA, Waldman AD. Incidental findings found in "healthy" volunteers during imaging performed for research: current legal and ethical implications. Br J Radiol. 2010 Jun;83(990):456-65. doi: 10.1259/bjr/15877332. Epub 2010 Mar 24. PMID 20335427
- [Derived] Dupriez F, Tollet J, Nely H, Steenebruggen F, Peyskens L, Marissiaux L, Germeau B, Collard A, Mordant C, Thoma M, Penaloza A, de Castro BR. Point-of-care ultrasound diagnostic accuracy for fecal impaction in the emergency department: a prospective study. Intern Emerg Med. 2025 Nov 3. doi: 10.1007/s11739-025-04150-8. Online ahead of print. PMID 41182496
- See also: Point of care ultrasound use by Registered Nurses and Nurse Practitioners in clinical practice: An integrative review — https://doi.org/10.1016/j.colegn.2020.10.002